CLINICAL TRIAL: NCT03241771
Title: Impact of Direct Outreach to Expand Access to Naloxone in the Context of Standing Orders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Denver Health and Hospital Authority (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CO-16-2405; 1R01DA042059-01 (NIH)
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Opioid Abuse; Overdose; Risk Behavior
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Risk-Taking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxone Navigator 1.0 (Experimental): Participants randomized to the Naloxone Navigator 1.0 arm will receive a link to the web-based resource. They will also receive usual care from their health plan, pharmacy and physicians. As part of usual care, participants will have access to naloxone through standing orders (i.e., they can request it without a prescription under their usual pharmacy benefit).
  Interventions: Behavioral: Naloxone Navigator 1.0
- Usual Care (No Intervention): Participants in the usual care arm will receive usual care from their health plan, pharmacy and physicians. As part of usual care, participants will have access to naloxone through standing orders (i.e., they can request it without a prescription under their usual pharmacy benefit).

INTERVENTIONS:
Behavioral: Naloxone Navigator 1.0 — Patients on chronic opioid therapy will be outreached via email, mail and phone. Within 1 month of enrollment into the trial, intervention participants will receive a link to the web-based resource to view. This is designed to provide overdose education, increase opioid risk awareness, and encourage patients to obtain naloxone.
  Other Names: Naloxone Navigator (NN)
  Arms: Naloxone Navigator 1.0

SUMMARY:
In the setting of naloxone standing orders, this study will assess if direct outreach with a web-based "Naloxone Navigator 1.0" to patients prescribed chronic opioid therapy (COT) changes opioid risk behaviors, increases naloxone uptake, and increases knowledge about overdose and naloxone

DETAILED DESCRIPTION:
This is a randomized study of a web-based naloxone educational resource (Naloxone Navigator 1.0) for adults prescribed chronic opioid therapy. This study will be conducted under new naloxone standing order legislation passed in Colorado. The Naloxone Navigator 1.0 will provide online training on how to recognize an opioid overdose and respond using naloxone. There will be two arms: one will receive a link to the Naloxone Navigator 1.0 and the other will receive usual care (no link). Outcomes will include opioid risk behavior, overdose and naloxone knowledge, naloxone dispensings, and overdose rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater prescribed chronic opioid therapy

Exclusion Criteria:

* Non-English speaking, hospice enrollment, do-not-resuscitate order, receipt of naloxone in the last 12 months, no internet access, not planning to continue to receive care in the same setting for the next 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Risk Behavior | 4 months
  Risk behavior will be assessed using the Opioid-Related Behaviors in Treatment (ORBIT) scale. The ORBIT is a brief scale used to identify recent risk behavior among patients receiving chronic opioid therapy.

SECONDARY OUTCOMES:
Patient Knowledge | Within 1 month of study enrollment
  Patient knowledge of overdose and naloxone will be measured using survey items adapted from the Opioid Overdose Knowledge Scale (OOKS). The OOKS is a scale measuring knowledge of overdose risks, warning signs, steps to address the overdose and appropriate use of naloxone.
Naloxone Dispensings | 4 months
  Electronic health records and pharmacy databases will be used to identify naloxone dispensings in the outpatient setting.
Opioid dose | 4 months
  We will calculate changes in the milligrams morphine equivalent dose
Drug Use Risk Behavior | 4 months
  Drug Use Risk Behavior will be assessed using the validated National Institutes on Drug Abuse-Modified (ASSIST) scale.
Alcohol Use Risk Behavior | 4 months
  Alcohol Use Risk Behavior will be assessed using the validated Alcohol Use Disorders Identification Test--Consumption (AUDIT-C Lite) scale. AUDIT-C Lite is a brief screener used to identify patients with alcohol use disorders or hazardous drinking behavior

OTHER OUTCOMES:
Pain Intensity | 4 months
  Pain intensity will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS Pain Intensity - Short Form instrument measures pain intensity over time
Overdose | 4 months
  Fatal and nonfatal overdoses will be assessed using International Classification of Disease (ICD)-10 codes in the electronic health record data and death records.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Binswanger, MD, Principal Investigator — Kaiser Permanente; Jason Glanz, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided